CLINICAL TRIAL: NCT05522101
Title: Mini-sized Magnetically Controlled Capsule Endoscopy vs. Normal-sized CE for Detection of Small Bowel in Children Under the Age of 10 Years：A Prospective，Multi-center，Randomized Controlled Trial
Brief Title: Mini-sized MCE for Detection of Small Bowel in Children Under the Age of 10 Years
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Shanghai Children's Hospital (Other); Xian Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Zhuan Liao, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Mini-sized MCE
Record Dates: First submitted 2022-08-04; First posted 2022-08-30 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Small Bowel Disease
Keywords: Children; Small Bowel Disease; Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mini-sized MCE (Experimental): AKES-31SW Capsule Endoscopy
  Interventions: Device: Mini-sized MCE
- Normal sized CE (Placebo Comparator): PillCam Capsule Endoscopy
  Interventions: Device: Normal-sized MCE

INTERVENTIONS:
Device: Mini-sized MCE — AKES-31SW capsule endoscopy（Mini-sized MCE), its diameter is 9.5mm, length is 24.5mm, weight is 3.0g, shooting frequency is 0.5-6fps, image resolution is 480*480, working time is not less than 8 hours. Mini-sized MCE is 0.6 times of traditional MCE in volume and weight, which is the smallest capsule in clinical application
  Arms: Mini-sized MCE
Device: Normal-sized MCE — Pillcam SB 3 capsule endoscopy（Normal-sized MCE), its diameter is 11.4mm, length is 26.2mm, weight is 3.0g, shooting frequency is 2-6fps, image resolution is 340*340, working time is not less than 8 hours.
  Arms: Normal sized CE

SUMMARY:
In this prospective randomized controlled trial, pediatric volunteers were enrolled and randomly underwent mini-sized MCE and normal-sized CE to compare the success rate of self-swallowing between mini-sized MCE and normal-sized CE during gastrointestinal examination.

DETAILED DESCRIPTION:
Magnetic controlled capsule endoscopy (MCE) is comparable to traditional gastroscopy (EGD) in the diagnosis of gastric diseases, and has been widely used in clinical practice. However, there are still some limitations in the application of MCE in digestive tract examination. Due to the large size of capsules at present, some patients have difficulty swallowing capsules during capsule swallowing, which leads to the failure of examination, and the proportion is higher in children patients. Therefore, in order to further improve the patient's comfort in swallowing capsules, our team developed a small MCE with a smaller size combined with innovation, which is 0.6 times of the conventional MCE in terms of volume and weight. This study aims to clarify the application efficacy of mini-MCE in gastrointestinal examination of adults and children through a multicenter clinical study comparing conventional capsule endoscopy with mini-magnetic-controlled capsule endoscopy. In order to ensure the efficacy of the capsule in the examination of digestive tract mucosa, and improve the ease of swallowing in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients and their legal guardians agreed to participate in the study and signed informed consent;
* 2 years ≤ age < 10 years;
* Pediatric patients with suspected small bowel disease who are scheduled for small bowel capsule endoscopy

Exclusion Criteria:

* Intestinal obstruction, stenosis, or fistula is known or suspected;
* Dysphagia or gastric emptying dysfunction;
* Severe asthma, dysphagia or gastroparesis and other emptying disorders;
* Known or suspected possibility of major bleeding from active digestive tract;
* The presence of a pacemaker in the body, except where the pacemaker is a new MRI-compatible product;
* Implanted cochlear implants, magnetic metal drug infusion pumps, nerve stimulators and other electronic devices, as well as magnetic metal foreign bodies;
* Those who plan to undergo magnetic resonance imaging (MRI) examination before capsule endoscopy discharge;
* Previous history of abdominal surgery affecting the normal structure of the digestive tract;
* Patients with mental illness;
* Allergic to macromolecular materials such as dimethyl silicone oil;
* Refuse to use electronic gastroscopy to deliver the capsule to the duodenum if the capsule cannot be swallowed by itself;
* Contraindications of intravenous anesthesia;
* Patients who have participated in or are participating in other clinical trials within three months;
* Any other factors considered by the investigator to be inappropriate for enrollment or to affect the participant's participation in the study.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 158 (Estimated)
Dates: Start 2022-10-20 (Estimated); Primary Completion 2023-07-20 (Estimated); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
Success rate of self-swallowing with Mini-sized MCE | 2 weeks
  Self-swallowing was defined as the subjects swallowing capsules for examination by themselves, and no endoscope or other instruments were needed to place capsules during the entire examination process

SECONDARY OUTCOMES:
Completion rate of capsule endoscopy gastric examination in two groups | 2 weeks
  The stomach was divided into six parts: cardia, fundus, body, antrum, angle and pylorus. The proportion of all subjects who completed complete observation of the six anatomical parts.
Completion rate of small bowel examination by capsule endoscopy in two groups | 2 weeks
  Small bowel examination completion definition: All subjects reached the cecum with capsule endoscopy and completed small bowel examination.
Success rate of instrument-assisted examination in the two groups | 2 weeks
  The success rate of device-assisted examination was defined as the proportion of small bowel examinations performed by endoscopists using endoscope-assisted capsules.
Two groups of capsule endoscopy swallowing time | 2 weeks
  Swallowing time was defined as the time between the time when the patient first placed the capsule in the mouth and the time when the patient took the first image of the esophagus.
Two groups of capsule endoscopy swallowing intake of water | 2 weeks
  Definition of water intake in swallowing capsule: The total amount of water ingested by the subject after swallowing the capsule successfully or unsuccessfully using a measuring cup.
The degree of difficulty of capsule swallowing in the two groups | 2 weeks
  Swallowing difficulty is assessed on a scale of 0-5, with 0 being no difficulty and 5 being the most difficult.
Factors affecting swallowing by capsule endoscopy | 2 weeks
  Physiological parameter such as BMI were recorded
Factors affecting gastrointestinal retention under capsule endoscopy | 2 weeks
  The incidence of capsule retention due to anesthesia or intestinal obstruction was recorded
The transmit time of esophagus, the transmit time of stomach, the transmit time of small intestine and the retention time of capsule in two groups | 2 weeks
  The time of the first esophageal image, the first stomach image, the first small intestine image, the first large intestine image and the last image taken by capsule endoscopy were recorded.
  Esophageal transmit time: time of first stomach image minus time of first esophageal image Stomach transmit time: time of first small intestine image minus time of first stomach image Small bowel transmit time: the time of the first large intestine image minus the time of the first small intestine image Total retention time of the capsule in vivo: total recording time of the capsule in vivo, which is the time of the last image of the capsule minus the time of the first image of the esophagus.
The time of gastric examination was magnetically controlled in the MCE group | 2 weeks
The rate of pylorus was magnetically controlled in the MCE group | 2 weeks
The detection rate of gastrointestinal lesions by capsule endoscopy in two groups | 2 weeks
Mucosal cleanliness of esophagus in two capsule endoscopy groups | 2 weeks
  Esophageal mucosa cleanliness score (Grade0: no bubbles, saliva or a small amount of bubbles, saliva, no impact on the observation of mucosa; Grade 1: moderate amount of bubbles and saliva, slight effect on observed mucosa; Grade 2: a large number of bubbles and saliva, which have a great influence on the observation of mucosa)
Mucosal cleanliness of stomach in two capsule endoscopy groups | 2 weeks
  Gastric mucosa cleanliness score:（Grade 1 : no adhesive mucus and foam, clear field of vision; Grade 2 : there is a small amount of mucus and foam, but the visual field is not blurred, which does not affect the integrity of the examination; Grade 3 : medium amount of mucus and foam, blurred visual field, affecting the integrity of the examination; Grade 4 : large amount of mucus and foam, blurred vision, affecting the integrity of the examination）
Mucosal cleanliness of small intestine in two capsule endoscopy groups | 2 weeks
  Small intestinal mucosa cleanliness score:
  Small bowel cleanliness score (Grade0: no fecal residue or a small amount of clear fluid, clear field of vision; Grade 1: There is a small amount of fecal residue or more clear liquid, and the visual field is still clear, which does not affect the observation; Grade 2: More fecal residue or turbid fecal fluid, blurred vision, affecting observation)
The integrity of esophageal mucosa was observed by capsule endoscopy in the two groups | 2 weeks
  Esophageal mucosal integrity The dentate line observation was evaluated mainly, including whether the dentate line could be observed, and the number of dentate line observation quadrants;
The integrity of gastric mucosa was observed by capsule endoscopy in the two groups | 2 weeks
  Gastric mucosa integrity assessment:
  The main anatomic sites such as cardia, fundus, body, Angle, antrum and pylorus were observed (grade 1: sufficient observation, ≥ 90% of gastric mucosa could be observed; Grade 2: Good observation, 70-90% of the gastric mucosa can be observed; Level 3: Insufficient observation, < 70% of gastric mucosa can be observed)
The integrity of small bowel mucosa was observed by capsule endoscopy in the two groups | 2 weeks
  The percentage of the total small bowel examination time in which the mucosa was clearly visible (> 50% visual field) was recorded
Incidence of adverse events | 2 weeks
  The rates of adverse events such as asphyxia by capsule aspiration, drug allergy and capsule retention were recorded
Overall inspection comfort score | 2 weeks
  A questionnaire survey was conducted on the overall comfort of Normal-sized CE and Mini-sized MCE, with 4 scores as very comfortable, 3 scores as comfortable, 2 scores as tolerable, 1 score as uncomfortable, and 0 score as very uncomfortable.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Principal Investigator — Changhai Hospital
Locations (4):
- China (4):
  - Qilu Children's Hospital, Jinan
  - Shanghai Changhai Hospital, Shanghai
  - Shanghai Children's Hospital, Shanghai
  - Xi'an Children's Hospital, Xi'an

IPD SHARING:
Plan to Share IPD: Yes
After finishing this study,We will make the data available to other researchers:including protocol,statistical analysis plan (SAP),informed consent form (ICF) and clinical study report (CSR).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 years
Access Criteria: The website of the journal where the results published,and ClinicalTrials.gov web site.

REFERENCES:
- [Background] Swaminath A, Legnani P, Kornbluth A. Video capsule endoscopy in inflammatory bowel disease: past, present, and future redux. Inflamm Bowel Dis. 2010 Jul;16(7):1254-62. doi: 10.1002/ibd.21220. PMID 20155845
- [Background] Arguelles-Arias F, Donat E, Fernandez-Urien I, Alberca F, Arguelles-Martin F, Martinez MJ, Molina M, Varea V, Herrerias-Gutierrez JM, Ribes-Koninckx C. Guideline for wireless capsule endoscopy in children and adolescents: A consensus document by the SEGHNP (Spanish Society for Pediatric Gastroenterology, Hepatology, and Nutrition) and the SEPD (Spanish Society for Digestive Diseases). Rev Esp Enferm Dig. 2015 Dec;107(12):714-31. doi: 10.17235/reed.2015.3921/2015. PMID 26671584
- [Background] Urs AN, Martinelli M, Rao P, Thomson MA. Diagnostic and therapeutic utility of double-balloon enteroscopy in children. J Pediatr Gastroenterol Nutr. 2014 Feb;58(2):204-12. doi: 10.1097/MPG.0000000000000192. PMID 24126830
- [Background] Gu Z, Wang Y, Lin K, Wang X, Cheng W, Wang L, Zhang T, Liu H. Magnetically Controlled Capsule Endoscopy in Children: A Single-center, Retrospective Cohort Study. J Pediatr Gastroenterol Nutr. 2019 Jul;69(1):13-17. doi: 10.1097/MPG.0000000000002292. PMID 30747810
- [Background] Cardey J, Le Gall C, Michaud L, Dabadie A, Talbotec C, Bellaiche M, Lamireau T, Mas E, Bridoux-Henno L, Viala J, Restier-Miron L, Lachaux A. Screening of esophageal varices in children using esophageal capsule endoscopy: a multicenter prospective study. Endoscopy. 2019 Jan;51(1):10-17. doi: 10.1055/a-0647-1709. Epub 2018 Sep 5. PMID 30184608
- [Background] Pai AK, Jonas MM, Fox VL. Esophageal Capsule Endoscopy in Children and Young Adults With Portal Hypertension. J Pediatr Gastroenterol Nutr. 2019 Dec;69(6):641-647. doi: 10.1097/MPG.0000000000002455. PMID 31365487
- [Background] Oliva S, Di Nardo G, Hassan C, Spada C, Aloi M, Ferrari F, Redler A, Costamagna G, Cucchiara S. Second-generation colon capsule endoscopy vs. colonoscopy in pediatric ulcerative colitis: a pilot study. Endoscopy. 2014 Jun;46(6):485-92. doi: 10.1055/s-0034-1365413. Epub 2014 Apr 28. PMID 24777427
- [Background] Xie M, Qian Y, Cheng S, Wang L, Shen R. Magnetically Guided Capsule Endoscopy in Pediatric Patients with Abdominal Pain. Gastroenterol Res Pract. 2019 May 8;2019:7172930. doi: 10.1155/2019/7172930. eCollection 2019. PMID 31205466
- [Background] Fritscher-Ravens A, Scherbakov P, Bufler P, Torroni F, Ruuska T, Nuutinen H, Thomson M, Tabbers M, Milla P. The feasibility of wireless capsule endoscopy in detecting small intestinal pathology in children under the age of 8 years: a multicentre European study. Gut. 2009 Nov;58(11):1467-72. doi: 10.1136/gut.2009.177774. Epub 2009 Jul 21. PMID 19625281
- [Background] Radhakrishnan C, Sefidani Forough A, Cichero JAY, Smyth HE, Raidhan A, Nissen LM, Steadman KJ. A Difficult Pill to Swallow: An Investigation of the Factors Associated with Medication Swallowing Difficulties. Patient Prefer Adherence. 2021 Jan 11;15:29-40. doi: 10.2147/PPA.S277238. eCollection 2021. PMID 33469272
- [Background] Ohmiya N, Oka S, Nakayama Y, Iwama I, Nakamura M, Shimizu H, Sumioka A, Abe N, Kudo T, Osawa S, Honma H, Okuhira T, Mtsufuji S, Imaeda H, Ota K, Matsuoka R, Hotta N, Inoue M, Nakaji K, Takamaru H, Ozeki K, Kobayashi T, Hosoe N, Tajiri H, Tanaka S. Safety and efficacy of the endoscopic delivery of capsule endoscopes in adult and pediatric patients: Multicenter Japanese study (AdvanCE-J study). Dig Endosc. 2022 Mar;34(3):543-552. doi: 10.1111/den.14104. Epub 2021 Sep 10. PMID 34379849
- [Background] Burgess CJ, McIntyre EC, Withers GD, Ee LC. Comparing swallowing of capsule to endoscopic placement of capsule endoscopy in children. JGH Open. 2017 Sep 18;1(1):11-14. doi: 10.1002/jgh3.12001. eCollection 2017 Sep. PMID 30483526
- [Background] Dan T, Dandan S, Enqiang L. Aspiration of a Magnetically Controlled Capsule Endoscopy. Gastroenterology. 2023 May;164(6):e30-e31. doi: 10.1053/j.gastro.2019.04.006. Epub 2019 Apr 11. No abstract available. PMID 30981792
- [Background] Melson J, Trikudanathan G, Abu Dayyeh BK, Bhutani MS, Chandrasekhara V, Jirapinyo P, Krishnan K, Kumta NA, Pannala R, Parsi MA, Sethi A, Trindade AJ, Watson RR, Maple JT, Lichtenstein DR. Video capsule endoscopy. Gastrointest Endosc. 2021 Apr;93(4):784-796. doi: 10.1016/j.gie.2020.12.001. Epub 2021 Feb 26. No abstract available. PMID 33642034
- [Background] Jiang B, Qian YY, Pan J, Jiang X, Wang YC, Zhu JH, Zou WB, Zhou W, Li ZS, Liao Z. Second-generation magnetically controlled capsule gastroscopy with improved image resolution and frame rate: a randomized controlled clinical trial (with video). Gastrointest Endosc. 2020 Jun;91(6):1379-1387. doi: 10.1016/j.gie.2020.01.027. Epub 2020 Jan 22. PMID 31981648
- [Background] Eliakim R. Where do I see minimally invasive endoscopy in 2020: clock is ticking. Ann Transl Med. 2017 May;5(9):202. doi: 10.21037/atm.2017.04.17. PMID 28567382
- [Background] Meltzer EO, Welch MJ, Ostrom NK. Pill swallowing ability and training in children 6 to 11 years of age. Clin Pediatr (Phila). 2006 Oct;45(8):725-33. doi: 10.1177/0009922806292786. PMID 16968958